CLINICAL TRIAL: NCT03849794
Title: The Effects of 4 Weeks of Chiropractic Care Plus Physiotherapy Compared to Physiotherapy Alone on Functional Outcomes in Chronic Stroke Patients: a Clinical Trial
Brief Title: Chiropractic Care Plus Physiotherapy Compared to Physiotherapy Alone in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Imran khan Niazi
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Chronic Stroke
Keywords: Chronic Stroke; Chiropractic Care; Physiotherapy
MeSH Terms: interventions — Physical Therapy Modalities; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the outcome assessors ( Physiotherapists), and data analysts will remain blinded to group allocation throughout the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Chiropractic Care Plus Physiotherapy
  Interventions: Other: Experimental Group
- Control group (Active Comparator): Physiotherapy
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental Group — Chiropractic Care A chiropractor will see participants in the experimental group about 3 times per week using a pragmatic approach for 4 weeks, and each session will be approximately 15-20 minutes in duration. The spinal adjustments performed in this study will be high-velocity, low-amplitude thrusts to the spine, pelvic joints, extremities or instrument-assisted adjustments
  Physiotherapy:
  Physiotherapists will see participants in each group 3 times per week for four weeks. Each session will be approximately 40 minutes in duration. Physiotherapy interventions are likely to include stretches and exercises, massage and mobilization as required.
  Other Names: Chiropractic Care Plus Physiotherapy
  Arms: Experimental group
Other: Control group — The control group will receive the same physiotherapy intervention as the experimental group at the same frequency of care. The control group will also attend three passive movement sessions with the chiropractor each week, primarily to minimise the psychological effect of the interaction with the chiropractor, but also to act as a physiological control. These passive movement sessions will be 15 minutes in duration.
  Other Names: Physiotherapy+sham Chiropractic
  Arms: Control group

SUMMARY:
The Investigator recently conducted a study in patients who had suffered from a stroke where it investigated whether similar findings are observed following a single session of chiropractic care.36 The key findings from this study was that in a group of chronic stroke patients, with lower limb muscle weakness, plantar flexion muscle strength increased on average by 64.6% following a chiropractic care session and the change in muscle strength appears to be modulated by cortical factors as opposed to modulation at the spinal level.

Based on the promising results of this initial study now planning to perform a pragmatic pilot clinical trial that will investigate the effects of 4 weeks of chiropractic care on clinical measures associated with stroke rehabilitation and function

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death and disability in the world. It is estimated that 17 million people per year suffer from a significant stroke worldwide, with 5 million of those people experiencing long term physical disability following the stroke. The global burden of stroke continues to rise even though the rate of stroke-related mortality has decreased over recent years. Stroke often results in prolonged physical, emotional, social and financial consequences for stroke survivors, family, friends, and caregivers. One of the most commonly occurring deficits associated with strokes is hemiparesis, which affects upper limb function, or an individual's ability to stand, balance or walk. The long term impaired nervous system function that accompanies many strokes means millions of stroke survivors around the world are reliant on care-givers to assist them with rudimentary activities of daily living such as bathing, dressing, and toileting. The burden of care is immense and has a significant impact on modern society.

This burden is even higher in developing countries. Disability-adjusted life years (DALYs), which is a measure of both years of life lost and years lived with a disability, is seven times higher in developing countries compared to high-income countries. While part of this difference is possibly due to differences in age, incidence, and mortality in developing countries; the mortality of stroke has dropped by 20% while the age-standardized incidence of stroke increased by 12% between 1990 and 2010 in low and middle-income countries. This means more people have strokes, more survive, and as a result, the burden of stroke is even greater in developing countries.

Numerous rehabilitative approaches have been shown to promote motor recovery after a stroke, but advanced strategies are constantly being developed and tested in an attempt to improve long term outcomes for stroke survivors. One possible intervention that may improve post-stroke motor recovery, but has to date not been adequately tested, is chiropractic care.

Over the past two decades, numerous research studies have shown that chiropractic care can significantly influence central neural function. Studies have shown changes in somatosensory processing, sensorimotor integration and motor control following as little as a single session of chiropractic care. Sensorimotor integration is the ability of the central nervous system (CNS) to integrate sensory information from different body parts and formulate appropriate motor outputs to muscles. Effective sensorimotor integration is essential when learning new motor skills, or recovering from an injury. Another essential component for accurate movement, learning new motor skills, and/or recovering from an injury is the accuracy of internal representations of our body map, or body schema. It is essential for our brain to be accurately aware of the location of our limbs and core body in 3D space. The spine is linked biomechanically and neurologically to the limbs and yet, it know very little about how altered sensory feedback from the spine affects limb sensorimotor integration and motor performance. However, there is emerging evidence that altered spinal sensory input can alter central neural processing, possibly by impacting the brains inner body schema. There is also emerging evidence that improving spinal function with chiropractic care can rapidly alter central neural function in a variety of ways, and that these changes outlast the altered changes of input, i.e. that they are neural plastic changes.

It has been hypothesised that the central neural plastic changes that are observed following chiropractic care may be due to improvements in spinal function associated with the correction of vertebral subluxations. Vertebral subluxations have been defined as a diminished state of being, comprising of a state of reduced coherence, altered biomechanical function, altered neurological function and altered adaptability.

If chiropractic care results in improvements in spinal function that have a central neural plastic effect, this may be important for a variety of clinical populations. Recently, groups reported an increase in lower limb muscle strength of 16% in reasonably healthy subjects following a single session of chiropractic care.Study also assessed possible neural plastic changes associated with spinal manipulation by assessing the H-reflex and V-waves. By also assessing these reflexes it helped to establish whether changes in strength following chiropractic adjustments were due to spinal or supraspinal influences. The H-reflex and V-waves are neurophysiological measures that have previously been shown to change following chiropractic care and are also important indicators of changes in central nervous system function that are important for motor recovery following a stroke. The H-reflex is largely modulated by presynaptic inhibition, and motoneuron excitability (spinal input), and the V-wave is a measure of supraspinal input, or cortical drive, to the motor neuron pool. It found changes in both the H-reflex and V-waves associated with increases in strength in our study.

Other small studies have also shown an increase in strength following a single session of chiropractic care. It also recently found a significant 8% increase in lower limb muscle strength in elite taekwondo athletes after a single session of chiropractic care. One previous controlled pilot study reported a significant increase in quadriceps muscle strength following a single chiropractic adjustment session. However group allocation was not randomised, which resulted in baseline group differences, and post-intervention between-group differences were not significant (p=0.2).It also reported a decrease in quadriceps muscle inhibition and increased quadriceps muscle activation following a chiropractic adjustment session. If these changes are lasting, and also occur in people who have suffered from a stroke, they may be important for stroke recovery.

The improvements in muscle strength and fatigue following chiropractic care observed in these studies are likely attributed to increased descending drive and/or modulation in synaptic efficacy of primary afferents or their connections at spinal cord level. This may have clinical implications for a variety of patient populations and in particular, people who have suffered from a stroke, who are likely to benefit from gains in power and strength if they occur following chiropractic care.

ELIGIBILITY:
Inclusion Criteria:

* patients must have suffered from a stroke at least 12 weeks prior to their involvement in the trial
* have ongoing neurological deficits
* upper and/or lower limb weakness
* with a Fugl-Meyer Assessment (FMA) motor score of less than 80 at the time of enrolment.

Exclusion Criteria:

* have absolute contraindications to chiropractic adjustments
* have experienced previous significant adverse reactions to chiropractic care or any type of manual therapy
* are unable to provide informed consent to participate in the trial due to cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | baseline,4th week, 8th week
  Changes from the Baseline, The Fugl-Meyer Assessment (FMA) (combined upper and lower limb )is a stroke-specific, performance-based impairment index. It is designed to assess motor function, balance, sensation and joint function in patients with post-stroke hemiplegia. It is applied clinically and in research to determine stroke severity, describe motor recovery, and to plan and assess treatment. Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. Only the Motor Part: Motor score: ranges from 0 (hemiplegia) to 100 points (normal motor performance).Classifications for impairment severity have been proposed based on FMA Total motor scores (out of 100 points) [< 50 = Severe, 50-84 = Marked, 85-94 = Moderate and 95-99 = Slight ]

SECONDARY OUTCOMES:
Stroke Specific Quality of Life Scale | baseline,4th week, 8th week
  Changes from the Baseline, The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life (HRQOL) specific to patients with stroke. Scoring: each item shall be scored with the following key Total help - Couldn't do it at all - Strongly agree (1), A lot of help - A lot of trouble - Moderately agree (2), Some help - Some trouble - Neither agree nor disagree (3), A little help - A little trouble - Moderately disagree (4) No help needed - No trouble at all - Strongly disagree (5)
Modified Rankin Scale (mRS) | baseline,4th week, 8th week
  Changes from the Baseline, The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
Timed up and Go Test (TUG) | baseline,4th week, 8th week
  Changes from the Baseline, The TUG is a widely used test of basic functional mobility that is sensitive to change and is suitable for the assessment of stroke patients.The TUG involves participants standing from a seated position, walking 3 meters, turning around and returning to sit in the chair. The time to complete this task is recorded using a stopwatch.
Heart Rate Variability(HRV) | baseline,4th week, 8th week
  HRV will be used as a objective assessment of psychological health and stress for the patients.
Daily Movement | 1 Week
  Accelerometer sensor will be used for a subset of patients to monitor the amount of daily movement during a week chosen randomly out of 4 weeks of care.
Blood Marker (Brain-derived neurotrophic factor, BDNF) | baseline,4th week, 8th week
  BDNF, is a protein that, in humans, is encoded by the BDNF Gene. BDNF is a member of the neurotrophin family of growth factors, which are related to the canonical nerve growth factor. Neurotrophic factors are found in the brain and the periphery. Changes from the baseline; BDNF levels were evaluated using immunoenzymatic method (ELISA) in plasma samples taken in each patient.
Blood marker (Glial cell-derived neurotrophic factor, GDNF) | baseline,4th week, 8th week
  Glial cell-derived neurotrophic factor (GDNF) is a protein that, in humans, is encoded by the GDNF gene. GDNF is a small protein that potently promotes the survival of many types of neurons. Changes from the baseline; GDNF levels were evaluated using immunoenzymatic method (ELISA) in plasma samples taken in each patient.
Blood Marker (Insulin-like growth factor 2, IGF2) | baseline,4th week, 8th week
  Insulin-like growth factor 2 is one of three protein hormones that share structural similarity to insulin. Changes from the baseline; IGF2 levels were evaluated using immunoenzymatic method (ELISA) in plasma samples taken in each patient.

OTHER OUTCOMES:
Transcranial Magnetic Stimulation (change in level of cortico-spinal cord excitability) | 1 Week
  TMS will be used in pre and post intervention in first session only for those patients for whom motor evoked response can be evoked at resting state.
  A TMS assessment involves applying consistent magnetic stimuli to the brain and recording EMG activity from the targeted muscle. The level of activity in the muscle will change based on the level of excitability in the nervous system. It will assess whether the level of excitability changes pre and post the different interventions that we will be applying based on the EMG recordings of the target muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherzai AZ, Elkind MS. Advances in stroke prevention. Ann N Y Acad Sci. 2015 Mar;1338:1-15. doi: 10.1111/nyas.12723. PMID 25779474
- [Background] Clarke DJ, Forster A. Improving post-stroke recovery: the role of the multidisciplinary health care team. J Multidiscip Healthc. 2015 Sep 22;8:433-42. doi: 10.2147/JMDH.S68764. eCollection 2015. PMID 26445548
- [Background] Bennett DA, Krishnamurthi RV, Barker-Collo S, Forouzanfar MH, Naghavi M, Connor M, Lawes CM, Moran AE, Anderson LM, Roth GA, Mensah GA, Ezzati M, Murray CJ, Feigin VL; Global Burden of Diseases, Injuries, and Risk Factors 2010 Study Stroke Expert Group. The global burden of ischemic stroke: findings of the GBD 2010 study. Glob Heart. 2014 Mar;9(1):107-12. doi: 10.1016/j.gheart.2014.01.001. PMID 25432120
- [Background] Chen JC, Shaw FZ. Progress in sensorimotor rehabilitative physical therapy programs for stroke patients. World J Clin Cases. 2014 Aug 16;2(8):316-26. doi: 10.12998/wjcc.v2.i8.316. PMID 25133141
- [Background] Feigin VL. Stroke in developing countries: can the epidemic be stopped and outcomes improved? Lancet Neurol. 2007 Feb;6(2):94-7. doi: 10.1016/S1474-4422(07)70007-8. No abstract available. PMID 17239789
- [Background] Krishnamurthi RV, Feigin VL, Forouzanfar MH, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson LM, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, Risk Factors Study 2010 (GBD 2010); GBD Stroke Experts Group. Global and regional burden of first-ever ischaemic and haemorrhagic stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet Glob Health. 2013 Nov;1(5):e259-81. doi: 10.1016/S2214-109X(13)70089-5. Epub 2013 Oct 24. PMID 25104492
- [Background] Veerbeek JM, Langbroek-Amersfoort AC, van Wegen EE, Meskers CG, Kwakkel G. Effects of Robot-Assisted Therapy for the Upper Limb After Stroke. Neurorehabil Neural Repair. 2017 Feb;31(2):107-121. doi: 10.1177/1545968316666957. Epub 2016 Sep 24. PMID 27597165
- [Background] Greisberger A, Aviv H, Garbade SF, Diermayr G. Clinical relevance of the effects of reach-to-grasp training using trunk restraint in individuals with hemiparesis poststroke: A systematic review. J Rehabil Med. 2016 Apr 28;48(5):405-16. doi: 10.2340/16501977-2077. PMID 27008369
- [Background] Wist S, Clivaz J, Sattelmayer M. Muscle strengthening for hemiparesis after stroke: A meta-analysis. Ann Phys Rehabil Med. 2016 Apr;59(2):114-24. doi: 10.1016/j.rehab.2016.02.001. Epub 2016 Mar 8. PMID 26969343
- [Background] Haavik H, Murphy B. Subclinical neck pain and the effects of cervical manipulation on elbow joint position sense. J Manipulative Physiol Ther. 2011 Feb;34(2):88-97. doi: 10.1016/j.jmpt.2010.12.009. PMID 21334540
- [Background] Haavik H, Murphy B. The role of spinal manipulation in addressing disordered sensorimotor integration and altered motor control. J Electromyogr Kinesiol. 2012 Oct;22(5):768-76. doi: 10.1016/j.jelekin.2012.02.012. Epub 2012 Apr 6. PMID 22483612
- [Background] Taylor HH, Murphy B. Altered central integration of dual somatosensory input after cervical spine manipulation. J Manipulative Physiol Ther. 2010 Mar-Apr;33(3):178-88. doi: 10.1016/j.jmpt.2010.01.005. PMID 20350670
- [Background] Niazi IK, Turker KS, Flavel S, Kinget M, Duehr J, Haavik H. Changes in H-reflex and V-waves following spinal manipulation. Exp Brain Res. 2015 Apr;233(4):1165-73. doi: 10.1007/s00221-014-4193-5. Epub 2015 Jan 13. PMID 25579661
- [Background] Kerzoncuf M, Bensoussan L, Delarque A, Durand J, Viton JM, Rossi-Durand C. Plastic changes in spinal synaptic transmission following botulinum toxin A in patients with post-stroke spasticity. J Rehabil Med. 2015 Nov;47(10):910-6. doi: 10.2340/16501977-2014. PMID 26424152
- [Background] Fimland MS, Moen PM, Hill T, Gjellesvik TI, Torhaug T, Helgerud J, Hoff J. Neuromuscular performance of paretic versus non-paretic plantar flexors after stroke. Eur J Appl Physiol. 2011 Dec;111(12):3041-9. doi: 10.1007/s00421-011-1934-z. Epub 2011 Apr 1. PMID 21455614
- [Background] Pandian S, Arya KN, Kumar D. Minimal clinically important difference of the lower-extremity fugl-meyer assessment in chronic-stroke. Top Stroke Rehabil. 2016 Aug;23(4):233-9. doi: 10.1179/1945511915Y.0000000003. Epub 2016 Apr 16. PMID 27086865
- [Background] Arya KN, Verma R, Garg RK. Estimating the minimal clinically important difference of an upper extremity recovery measure in subacute stroke patients. Top Stroke Rehabil. 2011 Oct;18 Suppl 1:599-610. doi: 10.1310/tsr18s01-599. PMID 22120029
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Derived] Holt K, Niazi IK, Amjad I, Kumari N, Rashid U, Duehr J, Navid MS, Shafique M, Haavik H. The Effects of 4 Weeks of Chiropractic Spinal Adjustments on Motor Function in People with Stroke: A Randomized Controlled Trial. Brain Sci. 2021 May 21;11(6):676. doi: 10.3390/brainsci11060676. PMID 34064209